CLINICAL TRIAL: NCT00820053
Title: Eastern Hepatobilliary Surgical Hospital
Brief Title: A Trial of Adjuvant Transarterial Chemoembolization (TACE) for Preventing Tumor Recurrence After Liver Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EHBH-RCT-2008-014-2
Record Dates: First submitted 2009-01-07; First posted 2009-01-09 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; adjuvant therapy; TACE; time to recurrence; overall survival
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Epirubicin; Ethiodized Oil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no adjuvant TACE (No Intervention): controll group with patients who don't receive any adjuvant therapy after liver resection, to compare with the treatment group with patients who receive adjuvant TACE after liver resection
- adjuvant TACE (Experimental): patients who adjuvant TACE after liver resection
  Interventions: Drug: epirubicin and lipiodol

INTERVENTIONS:
Drug: epirubicin and lipiodol — using the technology of Seldinger,The drugs (30 mg epirubicin mixed with 5 ml lipiodol) are given via hepatica propria artery.
  Other Names: transarterial chemoembolization
  Arms: adjuvant TACE

SUMMARY:
The aim of this study is to analyze the therapeutic effect of adjuvant TACE after resection.Patients receiving curative resection (R0) were randomized to postoperative TACE group and no TACE group. The time to recurrence ,the overall survival as well as the incidence of complications after therapy was observed to confirm the role of adjuvant TACE.

DETAILED DESCRIPTION:
Although resection of hepatocellular carcinoma is potentially curative, local recurrence is common with the recurrence rate higher than 50% during 5 years. So to reduce the recurrence rate of HCC, some interventions had been tried in clinic, including transarterial chemoembolization (TACE), immunotherapy, and interferon treatment etc. But few of these adjuvant therapies had been proved effective and their long term efficacy and clinical application remained further explored.

TACE had been prove to be effective in patients with advanced stage of HCC in randomized controlled trials and meta-analysis, but the role of adjuvant TACE after liver resection is controversial. The results getting from different randomized control trials varied significantly because of the bias of patient selection, different study design，the small size of sample, different drug used in chemotherapy and lack of proper stratification…,so a big sample size, well patients selected and well designed randomized controlled trial is needed to further confirm the role of the postoperative TACE.

Patients with HCC who received curative liver resection (R0) were randomly assigned 1:1 by the doctors to receive no adjuvant TACE(control group) or TACE(treatment group). All patients in the treatment group received adjuvant TACE 45 days after liver resection. The outcomes of patients were evaluated during the 3-years follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients > 18 years and <=70 years of age.
2. Patients with HCC who received curative liver resection (R0).
3. Criteria of liver function: Child A-B level, serum bilirubin ≤ 1.5 times the upper limit of normal value,alanine aminotransferase and aspartate aminotransferase ≤ 2 times the upper limit of normal value.
4. No dysfunction in major organs; Blood routine, kidney function, cardiac function and lung function are basically normal. Hb ≥90g/L,WBC ≥3.000 cells/mm³,platelets ≥80.000 cells/mm³ .
5. Karnofsky Performance Score performance over 60 .
6. Patients who can understand this trial and have signed information consent

Exclusion Criteria:

1. Patients with apparent cardiac, pulmonary, cerebronic and renal dysfunction,which may affect the treatment of liver cancer.
2. Patients with other diseases which may affect the treatment mentioned here.
3. Patients with medical history of other malignant tumors.
4. Subjects participating in other clinical trials.
5. Extrahepatic metastasis, portal vein or other major vascular involvement. liver function:Child C.
6. Patients would not sign the consent to the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2010

SECONDARY OUTCOMES:
Time to recurrence | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Shen feng, MD, Study Chair — Eastern hepatobilliary surgery hospital
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China